CLINICAL TRIAL: NCT01956552
Title: Changes in Phenotype and Genotype of Breast Cancers During the Metastatic Process and Optimization of Therapeutic Targeting
Brief Title: Changes in Phenotype and Genotype of Breast Cancers During the Metastatic Process and Optimization of Therapeutic Targeting (ESOPE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IC 2009-05
Record Dates: First submitted 2013-09-26; First posted 2013-10-08 (Estimated); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer; Tumor biopsy; Phenotype and genotype characterization
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: biopsy or cytopuncture

SUMMARY:
The primary objective is to compare the phenotype and genotype of the primary tumor with those of its metastases in order to optimize the treatment of metastatic disease, in patients presenting with first metastatic progression of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in the study, patients must fulfill all of the following criteria:

Female patients. Age ≥ 18 years. ECOG performance status ≤ 2. Metastatic breast carcinoma, either at diagnosis or at first metastatic relapse.

Available FFPE +/- frozen primary tumor samples. Evaluable metastatic disease. Metastatic disease outside any previous radiotherapy field (e.g. sub-clavicular or internal mammary lymph nodes).

Metastatic disease accessible to either percutaneous or surgical sampling. Signed written informed consent (approved by an Independent Ethics Committee and obtained prior to any study-specific screening procedure).

Social and psychological welfare in concordance with compliance to the study.

Exclusion Criteria:

To be eligible to participate in the study, patients must fulfill none of the following criteria:

Bilateral or multifocal breast cancer. Isolated local or contralateral relapse.

Solitary bone and/or brain metastatic disease unless :

Metastatic sites eligible for a therapeutic surgery. Metastatic sites sampled for diagnosis purpose. Past or current history of malignant neoplasms, except for curatively treated basal and squamous cell carcinoma of the skin. Carcinoma in situ of the cervix. Any coagulopathy contraindicating tumor biopsy. Presence of a contraindication to general anesthesia, if required.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2009-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
To assess the phenotype ant genotype discrepancies regarding hormonal receptor, FISH status and proliferation between the primary tumor and the first metastatic progression. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: SIGAL BRIGITTE, MD, Principal Investigator — Institut Curie
Locations (6):
- France (6):
  - Centre Oscar Lambret, Lille
  - Hopital Saint Louis, Paris
  - Institut Curie, Paris
  - Institut Curie HOPITAL RENE HUGUENIN, Saint-Cloud
  - INSTITUT DE CANCEROLOGIE DE L'OUEST René Gauducheau, Saint-Herblain
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Derived] Callens C, Driouch K, Boulai A, Tariq Z, Comte A, Berger F, Belin L, Bieche I, Servois V, Legoix P, Bernard V, Baulande S, Chemlali W, Bidard FC, Fourchotte V, Salomon AV, Brain E, Lidereau R, Bachelot T, Saghatchian M, Campone M, Giacchetti S, Zafrani BS, Cottu P. Molecular features of untreated breast cancer and initial metastatic event inform clinical decision-making and predict outcome: long-term results of ESOPE, a single-arm prospective multicenter study. Genome Med. 2021 Mar 15;13(1):44. doi: 10.1186/s13073-021-00862-6. PMID 33722295